CLINICAL TRIAL: NCT06312176
Title: An Open-label, Randomized Phase 3 Study of MK-2870 as a Single Agent and in Combination With Pembrolizumab Versus Treatment of Physician's Choice in Participants With HR+/HER2- Unresectable Locally Advanced or Metastatic Breast Cancer
Brief Title: A Study of Sacituzumab Tirumotecan (MK-2870) as a Single Agent and in Combination With Pembrolizumab (MK-3475) Versus Treatment of Physician's Choice in Participants With HR+/HER2- Unresectable Locally Advanced or Metastatic Breast Cancer (MK-2870-010)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2870-010; MK-2870-010 (Other: MSD); 2023-504918-29-00 (Registry Identifier: EU CT); U1111-1289-8119 (Registry Identifier: UTN); jRCT2031240476 (Registry Identifier: Japan Registry of Clinical Trials (jRCT))
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Breast Neoplasms
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1 (PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Breast Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Paclitaxel; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Capecitabine; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Sacituzumab tirumotecan (Experimental): Participants receive 4 mg/kg of sacituzumab tirumotecan once every 2 weeks (Q2W) via intravenous (IV) infusion until progressive disease or discontinuation.
  Interventions: Drug: Sacituzumab tirumotecan
- Arm B:Pembrolizumab + Sacituzumab tirumotecan (Experimental): Participants receive 4 mg/kg of sacituzumab tirumotecan Q2W via IV infusion until progressive disease or discontinuation PLUS 400 mg of pembrolizumab once every 6 weeks (Q6W) via IV infusion for up to 18 administrations (up to ~2 years).
  Interventions: Drug: Sacituzumab tirumotecan; Biological: Pembrolizumab
- Arm C: Treatment of Physician's Choice (TPC) (Active Comparator): At the physician's discretion, participants receive chemotherapy of 80 mg/m^2 of paclitaxel once every week (Q1W) via IV infusion OR 90 mg/m^2 of paclitaxel once every 4 weeks (Q4W) via IV infusion OR 100 mg/m^2 of nab-paclitaxel Q4W via IV infusion OR 1000 mg/m^2 of capecitabine every 3 weeks (Q3W) orally OR 50 mg/m^2 of liposomal doxorubicin once every 4 weeks (Q4W) via IV infusion, until progressive disease or discontinuation.
  Interventions: Drug: Paclitaxel; Drug: Nab-paclitaxel; Drug: Capecitabine; Drug: Liposomal doxorubicin

INTERVENTIONS:
Drug: Sacituzumab tirumotecan — IV infusion
  Other Names: MK-2870
  Arms: Arm A: Sacituzumab tirumotecan; Arm B:Pembrolizumab + Sacituzumab tirumotecan
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®
  Arms: Arm B:Pembrolizumab + Sacituzumab tirumotecan
Drug: Paclitaxel — IV infusion
  Other Names: TAXOL®
  Arms: Arm C: Treatment of Physician's Choice (TPC)
Drug: Nab-paclitaxel — IV infusion
  Other Names: ABRAXANE®
  Arms: Arm C: Treatment of Physician's Choice (TPC)
Drug: Capecitabine — oral tablet
  Other Names: XELODA®
  Arms: Arm C: Treatment of Physician's Choice (TPC)
Drug: Liposomal doxorubicin — IV infusion
  Other Names: DOXIL®
  Arms: Arm C: Treatment of Physician's Choice (TPC)

SUMMARY:
The purpose of this study is to compare sacituzumab tirumotecan as a single agent, and in combination with pembrolizumab, versus Treatment of Physician's Choice (TPC) in participants with hormone receptor positive/human epidermal growth factor receptor-2 negative (HR+/HER2-) unresectable locally advanced, or metastatic, breast cancer.

The primary hypotheses are that sacituzumab tirumotecan as a single agent and sacituzumab tirumotecan plus pembrolizumab are superior to TPC with respect to progression-free survival (PFS) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) by blinded independent central review (BICR) in all participants.

ELIGIBILITY:
Inclusion Criteria:

* Has unresectable locally advanced or metastatic centrally-confirmed hormone receptor positive (HR+)/human epidermal growth factor receptor 2 negative (HER2-) breast cancer
* Has radiographic disease progression on one or more lines of endocrine therapy for unresectable locally advanced/metastatic HR+/HER2- breast cancer, with one in combination with a CDK4/6 inhibitor
* Is a chemotherapy candidate
* Has an eastern cooperative oncology group (ECOG) performance status of 0 to 1 assessed within 7 days before randomization
* Has adequate organ function
* Human immunodeficiency virus (HIV)-infected participants must have well controlled HIV on antiretroviral therapy
* Participants who are Hepatitis B surface antigen (HBsAg) positive are eligible if they have received HBV antiviral therapy for at least 4 weeks, and have undetectable HBV viral load
* Participants with a history of Hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable

Exclusion Criteria:

* Has breast cancer amenable to treatment with curative intent
* Has experienced an early recurrence (<6 months after completing adjuvant/neoadjuvant chemotherapy) and therefore is eligible to receive second-line (2L) treatment
* Has symptomatic advanced/metastatic visceral spread at risk of rapidly evolving into life-threatening complications
* Has received prior chemotherapy for unresectable locally advanced or metastatic breast cancer
* Active autoimmune disease that has required systemic treatment in the past 2 years
* History of (noninfectious) pneumonitis/interstitial lung disease that requires steroids, or has current pneumonitis/interstitial lung disease
* Has an active infection requiring systemic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2024-04-14 (Actual); Primary Completion 2027-07-11 (Estimated); Study Completion 2031-04-12 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) ( sacituzumab tirumotecan versus treatment of physician's choice [TPC]; pembrolizumab + sacituzumab tirumotecan versus TPC) | Up to ~38 months
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first as assessed by Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1). PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by blinded independent central review (BICR) will be presented.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to ~77 months
  OS is defined as the time from randomization to death due to any cause.
Progression-Free Survival (PFS) (pembrolizumab + sacituzumab tirumotecan + versus sacituzumab tirumotecan) | Up to ~57 months
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first as assessed by Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1). PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. PFS as assessed by blinded independent central review (BICR) will be presented.
Objective Response Rate (ORR) | Up to ~57 months
  ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1). The percentage of participants who experience CR or PR as assessed by Blinded Independent Central Review (BICR) will be presented.
Duration of Response (DOR) | Up to ~57 months
  For participants who demonstrate a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1), DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR as assessed by Blinded Independent Central Review (BICR) will be presented.
Change from baseline in global health status/quality of life scores, on the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) | Baseline and up to ~77 months
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to the questions "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?" are scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better overall health status.
Change from baseline in physical functioning score, on the EORTC QLQ-C30 | Baseline and up to ~77 months
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to questions about their physical functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better level of physical functioning.
Change from baseline in emotional functioning score, on the EORTC QLQ-C30 | Baseline and up to ~77 months
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to questions about their emotional functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better level of emotional functioning.
Change from baseline in fatigue score, on the EORTC QLQ-C30 | Baseline and up to ~77 months
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to questions about their fatigue are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A lower score indicates a better level of function.
Change from baseline in diarrhea score, on the EORTC QLQ-C30 | Baseline and up to ~77 months
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to the question "Have you had diarrhea?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A lower score indicates a better level of function.
Time to first Deterioration (TTD) in global health status/quality of life scores, on the EORTC QLQ-C30 | Up to ~77 months
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to the questions "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?" are scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better overall health status. TTD is defined as the time from baseline to the first onset of a 10-point deterioration from baseline in global health status/quality of life combined score.
TTD in physical functioning score, on the EORTC QLQ-C30 | Up to ~77 months
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to questions about their physical functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better level of physical functioning. TTD is defined as the time from baseline to the first onset of a 10-point deterioration from baseline in the physical functioning score.
TTD in emotional functioning score, on the EORTC QLQ-C30 | Up to ~77 months
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to questions about their emotional functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better level of emotional functioning. TD is defined as the time from baseline to the first onset of a 10-point deterioration from baseline in the emotional functioning score.
TTD in fatigue score, on the EORTC QLQ-C30 | Up to ~77 months
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to questions about their fatigue are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A lower score indicates a better level of function. TTD is defined as the time from baseline to the first onset of a 10-point deterioration from baseline in the fatigue score.
TTD in diarrhea score, on the EORTC QLQ-C30 | Up to ~77 months
  The EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life of cancer patients. Participant responses to the question about their diarrhea are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A lower score indicates a better level of function. TTD is defined as the time from baseline to the first onset of a 10-point deterioration from baseline in the diarrhea score.
Number of participants who experience one or more adverse events (AEs) | Up to ~77 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of participants who discontinue study treatment due to an AE | Up to ~77 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (257):
- United States (45):
  - Ironwood Cancer & Research Centers ( Site 0066), Chandler, Arizona
  - Banner MD Anderson Cancer Center-Oncology ( Site 0004), Gilbert, Arizona
  - Providence Medical Foundation-Oncology ( Site 0020), Fullerton, California
  - Moores Cancer Center ( Site 0059), La Jolla, California
  - Cancer and Blood Specialty Clinic ( Site 0001), Los Alamitos, California
  - University of Colorado Anschutz Medical Campus ( Site 0061), Aurora, Colorado
  - UCHealth Cherry Creek Medical Center ( Site 0094), Denver, Colorado
  - University of Colorado Health - Highlands Ranch Hospital ( Site 0095), Highlands Ranch, Colorado
  - Yale Cancer Center ( Site 0060), New Haven, Connecticut
  - Stamford Hospital ( Site 0049), Stamford, Connecticut
  - AdventHealth Altamonte Springs ( Site 0021), Altamonte Springs, Florida
  - University of Florida College of Medicine ( Site 0063), Gainesville, Florida
  - Orlando Health Cancer Institute ( Site 0011), Orlando, Florida
  - Archbold Memorial Hospital-Lewis Hall Singletary Oncology Center ( Site 0032), Thomasville, Georgia
  - Rush University Medical Center ( Site 0079), Chicago, Illinois
  - University of Chicago Medical Center ( Site 0067), Chicago, Illinois
  - Saint Elizabeth Medical Center Edgewood-Cancer Care Center ( Site 0053), Edgewood, Kentucky
  - Mary Bird Perkins Cancer Center-Breast & GYN Pavilion ( Site 0042), Baton Rouge, Louisiana
  - Greenebaum Comprehensive Cancer Center ( Site 0036), Baltimore, Maryland
  - Mercy Medical Center - Baltimore-Medical Oncology and Hematology ( Site 0028), Baltimore, Maryland
  - Holy Cross Hospital ( Site 0073), Silver Spring, Maryland
  - Dana-Farber Cancer Institute-Breast Oncology Center ( Site 0037), Boston, Massachusetts
  - Henry Ford Health ( Site 0002), Detroit, Michigan
  - Saint Luke's Cancer Institute ( Site 0027), Kansas City, Missouri
  - Washington University School of Medicine ( Site 0076), St Louis, Missouri
  - NYU Langone Health - Brooklyn ( Site 0089), Brooklyn, New York
  - NYU Langone Hospital - Long Island ( Site 0090), Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center-Hematology and Oncology ( Site 0068), New York, New York
  - Hematology Oncology Associates of Rockland ( Site 0054), Nyack, New York
  - Stony Brook University-Cancer Center ( Site 0034), Stony Brook, New York
  - Levine Cancer Institute ( Site 0014), Charlotte, North Carolina
  - Zangmeister Cancer Center ( Site 7000), Columbus, Ohio
  - Providence Portland Medical Center ( Site 0044), Portland, Oregon
  - Providence St. Vincent Medical Center ( Site 0081), Portland, Oregon
  - Thomas Jefferson University - Clinical Research Institute ( Site 0056), Philadelphia, Pennsylvania
  - Texas Oncology-Dallas Presbyterian Hospital ( Site 8000), Dallas, Texas
  - UT Southwestern Medical Center ( Site 0050), Dallas, Texas
  - The Center for Cancer and Blood Disorders ( Site 0041), Fort Worth, Texas
  - Texas Oncology - San Antonio ( Site 8002), San Antonio, Texas
  - The University of Texas Health Science Center at Tyler dba UT Health East Texas HOPE Cancer Center ( Site 0057), Tyler, Texas
  - Inova Schar Cancer Institute ( Site 0025), Fairfax, Virginia
  - Bon Secours St. Francis Medical Center-Oncology Research ( Site 0015), Midlothian, Virginia
  - VCU Health Adult Outpatient Pavillion ( Site 0070), Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia (BRCC) ( Site 8001), Roanoke, Virginia
  - University Hospital and UW Health Clinics-Carbone Cancer Center ( Site 0040), Madison, Wisconsin
- Argentina (6):
  - Instituto Alexander Fleming-Alexander Fleming ( Site 0382), Buenos Aires, Buenos Aires F.D.
  - Fundacion Estudios Clinicos-Oncology ( Site 0384), Rosario, Santa Fe Province
  - Hospital Aleman-Oncology ( Site 0386), Buenos Aires
  - Centro de Educación Médica e Investigaciones clínicas "Dr. Norberto Quirno" (CEMIC) ( Site 0383), Buenos Aires
  - Hospital Italiano de Córdoba ( Site 0385), Córdoba
  - Fundación CORI para la Investigación y Prevención del Cáncer ( Site 0387), La Rioja
- Australia (4):
  - Macquarie University-MQ Health Clinical Trials Unit ( Site 2002), Macquarie University, New South Wales
  - Westmead Hospital ( Site 2000), Westmead, New South Wales
  - Frankston Hospital-Oncology and Haematology ( Site 2003), Frankston, Victoria
  - Fiona Stanley Hospital-Medical Oncology ( Site 2004), Murdoch, Western Australia
- Belgium (5):
  - Institut Jules Bordet-Medicine Oncology ( Site 1104), Anderlecht, Bruxelles-Capitale, Region de
  - Cliniques universitaires Saint-Luc-Medical Oncology ( Site 1103), Brussels, Bruxelles-Capitale, Region de
  - Jessa Ziekenhuis-Limburgs Oncologisch Centrum ( Site 1105), Hasselt, Limburg
  - AZ Maria Middelares-IKG ( Site 1106), Ghent, Oost-Vlaanderen
  - Université Catholique de Louvain-Namur - Centre Hospitalier -Oncology ( Site 1107), Namur
- Brazil (6):
  - Oncoclínica Oncologistas Associados-Clinical Research ( Site 0407), Teresina, Piauí
  - Hospital Moinhos de Vento ( Site 0403), Porto Alegre, Rio Grande do Sul
  - Hospital do Câncer Mãe de Deus ( Site 0404), Porto Alegre, Rio Grande do Sul
  - Instituto de Oncologia Saint Gallen ( Site 0412), Santa Cruz do Sul, Rio Grande do Sul
  - Instituto do Câncer Brasil - Unidade Taubaté ( Site 0408), Taubaté, São Paulo
  - IBCC - Núcleo de Pesquisa e Ensino ( Site 0401), São Paulo
- Canada (7):
  - BC Cancer Surrey ( Site 0315), Surrey, British Columbia
  - Southlake Health ( Site 0311), Newmarket, Ontario
  - Princess Margaret Cancer Centre ( Site 0310), Toronto, Ontario
  - CIUSSS de l'Est-de-l'Île-de-Montréal ( Site 0301), Montreal, Quebec
  - Jewish General Hospital ( Site 0303), Montreal, Quebec
  - CHU de Quebec Universite Laval - Hopital du Saint-Sacrement ( Site 0302), Québec, Quebec
  - Centre intégré de santé et de services sociaux du Bas Saint-Laurent- Hôpital régional de Rimouski ( Site 0308), Rimouski, Quebec
- Chile (6):
  - FALP-UIDO ( Site 0451), Santiago, Region M. de Santiago
  - Oncovida ( Site 0453), Santiago, Region M. de Santiago
  - Clínica RedSalud Vitacura ( Site 0455), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile ( Site 0454), Santiago, Region M. de Santiago
  - Bradfordhill ( Site 0452), Santiago, Region M. de Santiago
  - Bradford Hill Norte ( Site 0456), Antofagasta
- Colombia (5):
  - Fundacion Colombiana de Cancerología Clinica Vida ( Site 0506), Medellín, Antioquia
  - FUNDACION CTIC CENTRO DE TRATAMIENTO E INVESTIGACION SOBRE CANCER LUIS CARLOS SARMIENTO ANGULO ( Site 0507), Bogotá, Bogota D.C.
  - Sociedad De Oncología y Hematología Del Cesar SAS-Oncology ( Site 0501), Valledupar, Cesar Department
  - IMAT S.A.S ( Site 0502), Montería, Departamento de Córdoba
  - Fundación Valle del Lili ( Site 0508), Cali, Valle del Cauca Department
- Costa Rica (3):
  - CIMCA ( Site 0551), San José, Provincia de San José
  - Hospital Metropolitano - Sede Lindora ( Site 0550), Santa Ana, Provincia de San José
  - ICIMED ( Site 0552), San José
- Czechia (5):
  - Nemocnice Ceske Budejovice-Onkologicke oddeleni ( Site 1138), České Budějovice, Jihočeský kraj
  - Fakultni nemocnice Ostrava-Klinika onkologicka ( Site 1134), Ostrava-Poruba, Moravskoslezský kraj
  - Fakultni nemocnice Olomouc-Onkologicka klinika ( Site 1132), Olomouc, Olomoucký kraj
  - Fakultni nemocnice v Motole-Onkologicka klinika 2. LF UK a FN Motol ( Site 1136), Prague, Praha 5
  - Fakultni nemocnice Kralovske Vinohrady-Onkologická klinika ( Site 1135), Prague
- Denmark (5):
  - Rigshospitalet ( Site 1180), Copenhagen, Capital Region
  - Nordsjællands Hospital - Hillerød ( Site 1184), Hillerød, Capital Region
  - Næstved Sygehus ( Site 1182), Næstved, Region Sjælland
  - Odense Universitetshospital ( Site 1181), Odense, Region Syddanmark
  - Vejle Sygehus ( Site 1183), Vejle, Region Syddanmark
- France (7):
  - Hopital Prive Jean Mermoz-Oncology ( Site 1246), Lyon, Auvergne-Rhône-Alpes
  - Centre François Baclesse ( Site 1250), Caen, Calvados
  - Centre de Cancérologie du Grand Montpellier ( Site 1244), Montpellier, Languedoc-Roussillon
  - Hôpital privé du Confluent SAS-Service d'oncologie médicale ( Site 1242), Nantes, Loire-Atlantique
  - Pitie Salpetriere University Hospital ( Site 1249), Paris, Orne
  - Centre Hospitalier Universitaire de Poitiers-Pôle régional de cancérologie ( Site 1243), Poitiers, Vienne
  - Institut Curie-Oncology medical Department ( Site 1240), Paris
- Germany (8):
  - Universitaetsklinikum Erlangen-Klinik für Gynäkologie und Geburtshilfe ( Site 1301), Erlangen, Bavaria
  - Klinikum Ernst von Bergmann-Frauenklinik ( Site 1305), Potsdam, Brandenburg
  - Franziskus-Hospital Harderberg ( Site 1308), Georgsmarienhütte, Lower Saxony
  - Universitaetsklinikum Duesseldorf-Klinik für Frauenheilkunde & Geburtshilfe ( Site 1311), Düsseldorf, North Rhine-Westphalia
  - Kliniken Essen-Mitte, Evangelische Huyssens-Stiftung-Klinik für Senologie/ Brustzentrum ( Site 1300), Essen, North Rhine-Westphalia
  - CaritasKlinikum Saarbruecken St. Theresia ( Site 1304), Saarbrücken, Saarland
  - SRH Wald-Klinikum Gera-Zentrum für klinische Studien ( Site 1315), Gera, Thuringia
  - Helios Klinikum Berlin-Buch-Klinik für Gynäkologie und Geburtshilfe ( Site 1314), Berlin
- Greece (6):
  - Errikos Dunant Hospital Center ( Site 1348), Athens, Attica
  - Aretaieio Hospital Oncology Unit ( Site 1345), Athens, Attica
  - Hygeia Hospital ( Site 1346), Marousi, Attica
  - University General Hospital of Larissa ( Site 1343), Larissa, Thessaly
  - Agios Loukas Clinic ( Site 1347), Thessaloniki
  - European Interbalkan Medical Center ( Site 1341), Thessaloniki
- Hong Kong (2):
  - Queen Mary Hospital ( Site 2040), Hksar
  - Prince of Wales Hospital ( Site 2041), Shatin
- Hungary (6):
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ-Onkoterápiás Klinika ( Site 1379), Szeged, Csongrád megye
  - Somogy Vármegyei Kaposi Mór Oktató Kórház-Oncology center ( Site 1371), Kaposvár, Somogy County
  - Zala Vármegyei Szent Rafael Kórház-Onkológiai osztály ( Site 1372), Zalaegerszeg, Zala County
  - Semmelweis Egyetem-Belgyógyászati és Onkológiai Klinika ( Site 1381), Budapest
  - Budapesti Uzsoki Utcai Kórház-Onkoradiológiai Osztály ( Site 1373), Budapest
  - Debreceni Egyetem Klinikai Kozpont-Onkológiai Klinika ( Site 1375), Debrecen
- India (4):
  - Tata Memorial Hospital-Medical Oncology ( Site 2053), Mumbai, Maharashtra
  - Kokilaben Dhirubhai Ambani Hospital & Medical Research Institute-Centre for cancer ( Site 2056), Mumbai, Maharashtra
  - All India Institute of Medical Sciences ( Site 2051), New Delhi, National Capital Territory of Delhi
  - Rajiv Gandhi Cancer Institute And Research Centre-Department of Clinical Research ( Site 2052), New Delhi, National Capital Territory of Delhi
- Ireland (3):
  - Bon Secours Cork Hospital ( Site 1422), Cork
  - St. Vincent's University Hospital-Medical Oncology Research Department ( Site 1420), Dublin
  - Mater Misericordiae University Hospital-Clinical Trials Research Unit ( Site 1423), Dublin
- Israel (4):
  - Rambam Health Care Campus-Oncology Division ( Site 1452), Haifa
  - Hadassah Medical Center ( Site 1451), Jerusalem
  - Rabin Medical Center ( Site 1453), Petah Tikva
  - Sheba Medical Center ( Site 1450), Ramat Gan
- Italy (9):
  - IRCCS - Istituto Romagnolo per lo Studio dei Tumori (IRST) "Dino Amadori" ( Site 1480), Meldola, Forli-Cesena
  - CRO-IRCCS ( Site 1478), Aviano, Friuli Venezia Giulia
  - Fondazione IRCCS Istituto Nazionale dei Tumori-Struttura Complessa Oncologia Medica 1 ( Site 1472), Milan, Lombardy
  - Istituto Europeo di Oncologia IRCCS-Divisione di Senologia Medica ( Site 1475), Milan, Lombardy
  - Istituto Clinico Humanitas ( Site 1476), Rozzano, Milano
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola ( Site 1474), Bologna
  - Ospedale San Martino ( Site 1479), Genova
  - Ospedale San Raffaele-Oncologia Medica ( Site 1471), Milan
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore ( Site 1477), Roma
- Japan (24):
  - Nagoya City University Hospital ( Site 2474), Nagoya, Aichi-ken
  - National Cancer Center Hospital East ( Site 2463), Kashiwa, Chiba
  - Hokkaido University Hospital ( Site 2460), Sapporo, Hokkaido
  - Tokai University Hospital ( Site 2473), Isehara, Kanagawa
  - St. Marianna University Hospital ( Site 2465), Kawasaki, Kanagawa
  - Kitasato University Hospital ( Site 2471), Sagamihara, Kanagawa
  - Kanagawa Cancer Center ( Site 2472), Yokohama, Kanagawa
  - Mie University Hospital ( Site 2483), Tsu, Mie-ken
  - Tohoku University Hospital ( Site 2482), Sendai, Miyagi
  - The University of Osaka Hospital ( Site 2476), Suita, Osaka
  - Saitama Medical University International Medical Center ( Site 2462), Hidaka, Saitama
  - Juntendo University Hospital ( Site 2468), Bunkyo, Tokyo
  - Cancer Institute Hospital of JFCR ( Site 2464), Koto, Tokyo
  - Showa Medical University Hospital ( Site 2466), Shinagawa, Tokyo
  - Tokyo Medical University Hospital ( Site 2467), Shinjuku, Tokyo
  - National Center for Global Health and Medicine ( Site 2469), Shinjuku, Tokyo
  - Fukushima Medical University Hospital ( Site 2461), Fukushima
  - Gifu University Hospital ( Site 2486), Gifu
  - Hiroshima City Hiroshima Citizens Hospital ( Site 2478), Hiroshima
  - Social medical corporation Hakuaikai Sagara Hospital ( Site 2481), Kagoshima
  - Kumamoto University Hospital ( Site 2480), Kumamoto
  - Kyoto University Hospital ( Site 2475), Kyoto
  - Okayama University Hospital ( Site 2485), Okayama
  - Osaka Prefectural Hospital Organization Osaka International Cancer Institute ( Site 2477), Osaka
- Malaysia (3):
  - Hospital Sultan Ismail ( Site 2153), Johor Bahru, Johor
  - Sarawak General Hospital ( Site 2154), Kuching, Sarawak
  - Pantai Hospital Kuala Lumpur ( Site 2151), Kuala Lumpur
- Mexico (6):
  - CIO - Centro de Inmuno-Oncología de Occidente ( Site 0592), Guadalajara, Jalisco
  - Grupo Médico ASSET-Clinical Research ( Site 0596), Mexico City, Mexico City
  - Health Pharma Professional Research S.A. de C.V: ( Site 0598), Mexico City, Mexico City
  - INCAN-TUMORES MAMARIOS ( Site 0597), Mexico City, Mexico City
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez"-Servicio de Oncología ( Site 0590), Monterrey, Nuevo León
  - CENTRO MEDICO ZAMBRANO HELLION-Centro de Cáncer de Mama ( Site 0595), San Pedro Garza García, Nuevo León
- Netherlands (7):
  - Ziekenhuis Rijnstate-Rijnstate Centrum Oncologisch Onderzoek ( Site 1524), Arnhem, Gelderland
  - Maastricht UMC+-Medical Oncology ( Site 1522), Maastricht, Limburg
  - Amphia Ziekenhuis, locatie Breda Molengracht-oncologie ( Site 1523), Breda, North Brabant
  - Catharina Ziekenhuis ( Site 1526), Eindhoven, North Brabant
  - Nederlands Kanker Instituut - Antoni van Leeuwenhoek (NKI-AVL)-medical oncology ( Site 1520), Amsterdam, North Holland
  - Isala, locatie Zwolle ( Site 1525), Zwolle, Overijssel
  - Meander Medisch Centrum ( Site 1521), Amersfoort, Utrecht
- Auckland City Hospital ( Site 2031), Auckland, New Zealand
- Peru (4):
  - Clinica Vallesur - AUNA ( Site 0652), Arequipa, Ariqipa
  - Hospital Militar Central Luis Arias Schereiber ( Site 0651), Jesús María, Lima
  - Oncosalud ( Site 0650), Lima, Muni Metro de Lima
  - IPOR Instituto Peruano de Oncología & Radioterapia ( Site 0653), Lima
- Philippines (2):
  - Metro Davao Medical and Research Center ( Site 2202), Davao City, Davao Del Sur
  - ST. LUKE'S MEDICAL CENTER-Medicine ( Site 2200), Quezon City, National Capital Region
- Poland (11):
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka-Ambulatorium Chemioterapii ( Site 1582), Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Mazowiecki Szpital Wojewódzki w Siedlcach-Siedleckie Centrum Onkologii ( Site 1584), Siedlce, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Klinika Nowotworów Piersi i Chirurgii ( Site 1580), Warsaw, Masovian Voivodeship
  - Mazowiecki Szpital Onkologiczny ( Site 1581), Wieliszew, Masovian Voivodeship
  - Mrukmed-Mrukmed ( Site 1592), Rzeszów, Podkarpackie Voivodeship
  - Bialostockie Centrum Onkologii ( Site 1585), Bialystok, Podlaskie Voivodeship
  - Szpitale Pomorskie Sp. z o. o.-Oddział Onkologii Klinicznej ( Site 1593), Gdynia, Pomeranian Voivodeship
  - Narodowy Instytut Onkologii - Oddzial w Gliwicach-Centrum Diagnostyki i Leczenia Chorob Piersi ( Site 1590), Gliwice, Silesian Voivodeship
  - Szpital Wojewódzki w Koszalinie. ( Site 1583), Poland, West Pomeranian Voivodeship
  - Zachodniopomorskie Centrum Onkologii ( Site 1588), Szczecin, West Pomeranian Voivodeship
  - Swietokrzyskie Centrum Onkologii, Samodzielny Publiczny Zakl-Klinika Onkologii Klinicznej, Dzial Ch ( Site 1595), Kielce, Świętokrzyskie Voivodeship
- Portugal (3):
  - Unidade Local de Saude Amadora/Sintra - Hospital Prof Dr Fernando Fonseca ( Site 1663), Lisbon, Lisbon District
  - Unidade Local de Saude de Santa Maria - Hospital de Santa Maria ( Site 1661), Lisbon
  - Instituto Português de Oncologia do Porto Francisco Gentil, EPE ( Site 1662), Porto
- Puerto Rico (2):
  - Puerto Rico Medical Research Center LLC ( Site 0675), Hato Rey
  - UPR Comprehensive Cancer Center-Comprehensive Cancer Center Hospital ( Site 0677), San Juan
- Romania (4):
  - Spitalul Clinic Filantropia ( Site 1703), Bucharest, București
  - SC Radiotherapy Center Cluj SRL-Oncologie Medicala ( Site 1702), Florești, Cluj
  - Centrul Medical Neolife- Baneasa ( Site 1704), Bucharest
  - Institutul Oncologic Cluj ( Site 1701), Cluj-Napoca
- Singapore (2):
  - National University Hospital ( Site 2250), Singapore, Central Singapore
  - Mount Alvernia ICON Cancer Center ( Site 2251), Singapore, North East
- South Africa (5):
  - CANCERCARE LANGENHOVEN DRIVE ONCOLOGY CENTRE ( Site 2905), Port Elizabeth, Eastern Cape
  - Wits Clinical Research ( Site 2903), Johannesburg, Gauteng
  - Curo Oncology ( Site 2908), Pretoria, Gauteng
  - Sandton Oncology Medical Group (Pty) Ltd ( Site 2911), Sandton, Gauteng
  - Cancercare Rondebosch Oncology-Clinical trials ( Site 2904), Cape Town, Western Cape
- South Korea (4):
  - Seoul National University Hospital-Internal Medicine ( Site 2353), Seoul
  - Severance Hospital, Yonsei University Health System-Medical oncology ( Site 2350), Seoul
  - Asan Medical Center-Department of Oncology ( Site 2352), Seoul
  - Samsung Medical Center-Division of Hematology/Oncology ( Site 2351), Seoul
- Spain (7):
  - HOSPITAL UNIVERSITARIO QUIRONSALUD MADRID ( Site 1758), Pozuelo de Alarcón, Madrid
  - HOSPITAL CLINICO DE VALENCIA-Oncology ( Site 1752), Valencia, Valenciana, Comunitat
  - Hospital Universitari Vall d'Hebron-Oncology ( Site 1750), Barcelona
  - Hospital Universitario Reina Sofia-Oncologia Medica ( Site 1754), Córdoba
  - Hospital Beata María Ana-oncology ( Site 1755), Madrid
  - HOSPITAL GENERAL UNIVERSITARIO GREGORIO MARAÑON-ONCOLOGY ( Site 1756), Madrid
  - Hospital Universitario Virgen Macarena ( Site 1757), Seville
- Sweden (3):
  - Karolinska Universitetssjukhuset Solna ( Site 1801), Stockholm, Stockholm County
  - Akademiska sjukhuset ( Site 1802), Uppsala, Uppsala County
  - Södra Älvsborgs Sjukhus Borås ( Site 1803), Borås, Västra Götaland County
- Switzerland (3):
  - University Hospital Basel-Gynecology & Gynecologic Oncology ( Site 1844), Basel, Canton of Basel-City
  - Spital Thun ( Site 1840), Thun, Canton of Bern
  - Brust-Zentrum ( Site 1841), Zurich, Canton of Zurich
- Taiwan (6):
  - Changhua Christian Hospital ( Site 2410), Changhua
  - Chang Gung Memorial Hospital at Kaohsiung-Oncology and Hematology ( Site 2413), Kaohsiung City
  - National Cheng Kung University Hospital-Surgery ( Site 2411), Tainan
  - National Taiwan University Hospital-Oncology ( Site 2415), Taipei
  - Mackay Memorial Hospital ( Site 2412), Taipei
  - Chang Gung Medical Foundation-Linkou Branch-General Surgery ( Site 2414), Taoyuan District
- Turkey (Türkiye) (8):
  - Dr. Abdurrahman Yurtaslan Ankara Onkoloji Egitim ve Arastırma Hastanesi ( Site 1878), Yenimahalle, Ankara
  - Medipol Mega Universite Hastanesi-oncology ( Site 1875), Stanbul, Istanbul
  - Adana Medical Park Seyhan Hastanesi-Medikal Onkoloji ( Site 1876), Adana
  - Hacettepe Universite Hastaneleri-oncology hospital ( Site 1870), Ankara
  - Memorial Ankara Hastanesi-Medical Oncology ( Site 1874), Ankara
  - Ankara Bilkent Şehir Hastanesi-Medical Oncology ( Site 1871), Ankara
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi-oncology ( Site 1872), Istanbul
  - Samsun Medical Park Hastanesi-medical oncology ( Site 1873), Samsun
- United Kingdom (6):
  - North West Cancer Centre ( Site 1944), Londonderry, Derry and Strabane
  - The Royal Cornwall Hospital ( Site 1943), Truro, England
  - St Bartholomew's Hospital-Centre for Experimental Cancer Medicine ( Site 1940), London, London, City of
  - University College London Hospital-Cancer Clinical Trials Unit ( Site 1942), London, London, City of
  - Blackpool Victoria Hospital ( Site 1941), Blackpool
  - City Hospital, Nottingham University Hospitals NHS Trust ( Site 1945), Nottingham

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26170&tenant=MT_MSD_9011